CLINICAL TRIAL: NCT02744339
Title: Evaluation of the Pharmacodynamic Effects of Riociguat in Subjects With Pulmonary Hypertension and Heart Failure With Preserved Ejection Fraction in a Randomized, Double Blind, Placebo Controlled, Parallel Group, Multicenter Study
Brief Title: Pharmacodynamic Effects of Riociguat in Pulmonary Hypertension and Heart Failure With Preserved Ejection Fraction
Acronym: DYNAMIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, DBonderman, Assoc.Prof.Priv.Doz.Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RIO-40400; 2014-003055-60 (EudraCT Number)
Record Dates: First submitted 2016-03-18; First posted 2016-04-20 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Hypertension, Pulmonary; Heart Failure With Normal Ejection Fraction
Keywords: PH-HFpEF
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — riociguat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Riociguat (Experimental): Riociguat up-titrated to a maximum of 1.5mg TID
  Interventions: Drug: Riociguat
- Placebo (Placebo Comparator): Placebo sham-titrated TID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Riociguat — Adempas up-titrated to max. 1.5mg TID
  Other Names: Adempas
  Arms: Riociguat
Drug: Placebo — Placebo sham-titrated TID
  Arms: Placebo

SUMMARY:
The primary objective of this study is to

• Assess the pharmacodynamic profile of riociguat in subjects with symptomatic pulmonary hypertension and heart failure with preserved ejection fraction

The secondary objectives of this study are to

* Assess safety and tolerability of riociguat in this study population
* Assess changes in dimensions of left and right ventricles and cardiac function parameters using cardiac magnetic resonance imaging

ELIGIBILITY:
Inclusion Criteria:

* 18 to <80 years of age at the time of informed consent (The lower age limit may be higher if legally required in participating countries.)
* Male and female subjects with symptomatic PH and HF-PEF (group 2 / 2.2 of Dana Point classification(4) and WHO class II to IV) (Other groups of PH, especially HF-REF, PAH, CTEPH, must have been ruled out according to accepted diagnostic procedures and guidelines, see section 5.1.2 Exclusion criteria.)
* PH-HF-PEF defined as:

  * LVEF ≥50%, diagnosed by echocardiography or left heart catheterization (LHC) within 30 days before randomization
  * PAPmean ≥25 mmHg at rest, measured by RHC
  * PAWP >15 mmHg at rest, measured by RHC
* Optimized therapy for hypertension
* The dose regimen of the background treatment must have been stable for >30 days before randomization. Diuretic therapy must have been stable for ≥1 week.
* RHC results for the definite diagnosis of PH not older than 12 weeks at Visit 1. RHC must have been performed in the participating center under standardized conditions
* CMRI must be performed at Visit 1 (baseline) or must not be older than 12 weeks with all parameters measured as listed in Section 7.3.3
* Women are eligible if not of childbearing potential, defined as:
* Postmenopausal women (i.e. last menstrual bleeding at least 2 years before randomization)
* Women with bilateral tubal ligation
* Women with bilateral ovariectomy
* Women with hysterectomy or, if of childbearing potential, women are eligible if
* A serum pregnancy test is negative at the pre-study visit, and The woman uses a combination of condoms and a safe and highly effective contraception method (hormonal contraception with implants or combined oral contraceptives, certain intrauterine devices) for the entire duration of the study.
* Able to understand and follow instructions and to participate in the study for its entire duration
* Written informed consent

Exclusion Criteria:

* PH in groups other than group 2.2 according to Dana Point classification.(4) In particular, PAH, CTEPH, and HF-REF must have been ruled out according to accepted diagnostic procedures and guidelines.
* Cardiac decompensation, with hospitalization or visit to the emergency department,

  ≤30 days before randomization
* Left heart disease because of to ischemic heart disease or dilated cardiomyopathy
* Resynchronization therapy at any time
* Need for intravenous (IV) diuretics ≤30 days before randomization
* Treatment with inotropes or IV vasodilators ≤30 days before randomization
* Pre-treatment with endothelin receptor antagonists (ERAs), phosphodiesterase type 5 (PDE5) inhibitors, or prostanoids ≤30 days before randomization, or with nitrates ≤7 days before randomization
* Subjects who medically require treatment with drugs that are not in line with the in- or exclusion criteria of this study or that are prohibited concomitant medications (see section 6.9) for this study
* Bronchial asthma or chronic obstructive pulmonary disease (COPD) with forced expiratory volume in 1 second (FEV1) <60% of predicted
* Restrictive lung disease with total lung capacity (TLC) <60% of predicted
* Subjects on oxygen therapy
* Severe congenital abnormalities of the lung, thorax, or diaphragm
* Clinically relevant hepatic dysfunction shown by:
* Aspartate aminotransferase (AST) ≥3 times the upper limit of normal (ULN) or
* Child Pugh stage B and C in cirrhotic subjects
* Severe renal impairment (glomerular filtration rate [GFR] <30mL/min/1.73 m2 calculated by the Modification of Diet in Renal Disease [MDRD] formula)
* Uncontrolled arterial hypertension (SBP >180 mmHg or diastolic blood pressure [DBP] >110 mmHg)
* SBP <110 mmHg at baseline
* Myocardial disease, such as ischemic or dilative infiltrative myocardial disease (i.e. amyloidosis, hypertrophic cardiomyopathy)
* Severe aortic or mitral stenosis, or any such stenosis with indication for surgery
* Coronary artery disease with angina of Canadian Cardiovascular Society (CCS) class III or IV or requiring nitrates, unstable angina, or acute myocardial infarction <90 days before randomization
* Reperfusion procedure (percutaneous coronary intervention [PCI] or coronary artery bypass graft [CABG]) <90 days before randomization, or <21 days in case of a negative stress test effect after PCI
* Stroke with persistent neurological deficit
* Subjects positive for human immunodeficiency virus (HIV)
* Resting HR while awake of <50 beats per minute (BPM) or >105 BPM (in case of atrial fibrillation >110 BPM)
* Participation in another clinical study <90 days before randomization
* Subjects with a medical disorder, condition, or history thereof that in the opinion of the investigator would impair the subject's ability to participate or complete the 26-week study
* Subjects with underlying medical disorders with an anticipated life expectancy below 2 years because of a non-cardiac disease (e.g. active cancer disease with localized and / or metastasized tumor mass)
* Subjects with a history of multiple drug allergies
* Subjects with hypersensitivity to the investigational drug or any of the excipients
* Previous assignment to treatment during this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline of cardiac output at rest, measured by right heart catheterization | Baseline and 26 weeks after study drug treatment
  Change from baseline of cardiac output at rest, measured by right heart catheterization after 26 weeks of study drug treatment

SECONDARY OUTCOMES:
Change from baseline in cardiac magnetic resonance imaging parameters | Baseline and 26 weeks after study drug treatment
  Change from baseline in right ventricular ejection fraction by cardiac magnetic resonance imaging
Change from baseline in cardiac magnetic resonance imaging parameters | Baseline and 26 weeks after study drug treatment
  Change from baseline in right ventricular volume by cardiac magnetic resonance imaging
Change from baseline in cardiac magnetic resonance imaging parameters | Baseline and 26 weeks after study drug treatment
  Change from baseline in left atrial area by cardiac magnetic resonance imaging
Change from baseline in cardiac magnetic resonance imaging parameters | Baseline and 26 weeks after study drug treatment
  Change from baseline in right atrial area by cardiac magnetic resonance imaging
Change from baseline in hemodynamic parameters other than cardiac output | Baseline and 26 weeks after study drug treatment
  Change from baseline in pulmonary vascular resistance by right heart catheterization
Change from baseline in hemodynamic parameters other than cardiac output | Baseline and 26 weeks after study drug treatment
  Change from baseline in pulmonary arterial wedge pressure by right heart catheterization
Change from baseline in hemodynamic parameters other than cardiac output | Baseline and 26 weeks after study drug treatment
  Change from baseline in transpulmonary gradient by right heart catheterization
Change from baseline in hemodynamic parameters other than cardiac output | Baseline and 26 weeks after study drug treatment
  Change from baseline in systemic vascular resistance by right heart catheterization
Change from baseline in WHO functional class | Baseline and 26 weeks after study drug treatment
Change from baseline in biomarker levels | Baseline and 26 weeks after study drug treatment
  Change from baseline in serum N-terminal prohormone B-type natriuretic peptide (NTproBNP)

OTHER OUTCOMES:
Change from baseline in T1-mapping parameters by CMR | Baseline and 26 weeks after study drug treatment
  Change from baseline in native T1 times of the left ventricular myocardium
Change from baseline in T1-mapping parameters by CMR | Baseline and 26 weeks after study drug treatment
  Change from baseline in extracellular volume of the left ventricular myocardium
Change from baseline in echocardiography parameters | Baseline and 26 weeks after study drug treatment
  Change from baseline in left ventricular end-systolic volume by echocardiography
Change from baseline in echocardiography parameters | Baseline and 26 weeks after study drug treatment
  Change from baseline in left ventricular end-diastolic volume by echocardiography
Change from baseline in echocardiography parameters | Baseline and 26 weeks after study drug treatment
  Change from baseline in tricuspid annular plan systolic excursion by echocardiography
Change from baseline in echocardiography parameters | Baseline and 26 weeks after study drug treatment
  Change from baseline in pressure gradient of tricuspid valve by echocardiography
Change from baseline in echocardiography parameters | Baseline and 26 weeks after study drug treatment
  Change from baseline in diameter of inferior vena cava by echocardiography
Change from baseline in echocardiography parameters | Baseline and 26 weeks after study drug treatment
  Change from baseline in respiratory collapsibility of inferior vena cava by echocardiography
Change from baseline in echocardiography parameters | Baseline and 26 weeks after study drug treatment
  Change from baseline in mitral peak velocity of early (E) filling by echocardiography
Change from baseline in echocardiography parameters | Baseline and 26 weeks after study drug treatment
  Change from baseline in mitral peak velocity of late (A) filling by echocardiography
Change from baseline in echocardiography parameters | Baseline and 26 weeks after study drug treatment
  Change from baseline in E-wave deceleration time by echocardiography
Change from baseline in echocardiography parameters | Baseline and 26 weeks after study drug treatment
  Change from baseline in left ventricular ejection fraction by echocardiography
Change from baseline in echocardiography parameters | Baseline and 26 weeks after study drug treatment
  Change from baseline in estimate of mean right atrial pressure by echocardiography
Change from baseline in echocardiography parameters | Baseline and 26 weeks after study drug treatment
  Change from baseline in systolic pulmonary artery pressure by echocardiography
Change from baseline in echocardiography parameters | Baseline and 26 weeks after study drug treatment
  Change from baseline in E/A ratio by echocardiography
Change from baseline in exercise capacity: 6-minute walk distance | Baseline and 26 weeks after study drug treatment
Change from baseline in exercise capacity: Borg CR 10 scale | Baseline and 26 weeks after study drug treatment
Change from baseline in quality of life scores: EQ-5D | Baseline and 26 weeks after study drug treatment
Change from baseline in quality of life scores: MLHF | Baseline and 26 weeks after study drug treatment
Events of special interest | Baseline and 26 weeks after study drug treatment
  Events of special interest considered for calculation of the combined endpoint "time to clinical worsening"
All-cause mortality | Baseline and 26 weeks after study drug treatment
Composite endpoint | Baseline and 26 weeks after study drug treatment
  Composite endpoint as defined by: time to death from cardiovascular causes or first hospitalization for a cardiovascular event, including acute or worsening heart failure, acute myocardial infarction, stroke, or ventricular arrhythmia

CONTACTS AND LOCATIONS:
Overall Officials: Diana Bonderman, MD, Principal Investigator — Medical University of Vienna; Johannes Kastner, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria